CLINICAL TRIAL: NCT02510794
Title: A Phase II, Multicenter, Randomized, Active Treatment-Controlled Study of the Efficacy and Safety of the Ranibizumab Port Delivery System for Sustained Delivery of Ranibizumab in Patients With Subfoveal Neovascular Age-Related Macular Degeneration
Brief Title: Study of the Efficacy and Safety of the Ranibizumab Port Delivery System for Sustained Delivery of Ranibizumab in Patients With Subfoveal Neovascular Age-Related Macular Degeneration
Acronym: LADDER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX28228
Record Dates: First submitted 2015-07-17; First posted 2015-07-29 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Port Delivery System with Ranibizumab 10mg/mL (Experimental): Participants had the Implant (prefilled with approximately 20 μL of 10-mg/mL ,approximately 0.2 mg dose, of ranibizumab) surgically inserted in the study eye at the Day 1 visit following their randomization visit. Starting at the Month 1 visit, participants were evaluated monthly for the need for Implant refill with the 10-mg/mL formulation of ranibizumab according to their randomization as per protocol-specified refill criteria.
  Interventions: Drug: Ranibizumab
- Port Delivery System with Ranibizumab 40mg/mL (Experimental): Participants had the Implant (prefilled with approximately 20 μL of 40-mg/mL, approximately 0.8 mg dose, of ranibizumab) surgically inserted in the study eye at the Day 1 visit following their randomization visit. Starting at the Month 1 visit, participants were evaluated monthly for the need for Implant refill with the 40-mg/mL formulation of ranibizumab according to their randomization as per protocol-specified refill criteria.
  Interventions: Drug: Ranibizumab
- Port Delivery System with Ranibizumab 100mg/mL (Experimental): Participants had the Implant (prefilled with approximately 20 μL of 100-mg/mL, approximately 2 mg dose, of ranibizumab) surgically inserted in the study eye at the Day 1 visit following their randomization visit. Starting at the Month 1 visit, participants were evaluated monthly for the need for Implant refill with the 100-mg/mL formulation of ranibizumab according to their randomization as per protocol-specified refill criteria.
  Interventions: Drug: Ranibizumab
- Intravitreal Injection with Ranibizumab 0.5mg (Active Comparator): Participants received ranibizumab 0.5 mg monthly ITV injections of 10 mg/mL formulation at Day 1 and every month thereafter.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab will be administered at dose of 0.5 mg monthly ITV injections of 10-mg/mL formulation or delivered through the implant with three different formulations.
  Other Names: Lucentis®

SUMMARY:
This is a Phase II multicenter, dose-ranging, randomized, active treatment (monthly ITV injection)-controlled study to evaluate the efficacy, safety, and pharmacokinetics of ranibizumab delivered through the Implant using three ranibizumab formulation arms (10 mg/mL, 40 mg/mL, and 100 mg/mL) compared with the control arm (0.5-mg monthly ITV injections of 10-mg/mL formulation) in participants with subfoveal neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with wet AMD within 9 months of screening visit
* Participant must have received at least 2 prior ITV anti-vascular endothelial growth factor (VEGF) injections. However, the most recent anti-VEGF injection must have been ranibizumab and must have occurred at least 7 days prior to the screening visit
* Demonstrated response to prior ITV anti-VEGF treatment
* Best Corrected Visual Acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) charts of 20/20-20/200 Snellen equivalent

Exclusion Criteria:

* Treatment with ITV anti-VEGF agents other than ranibizumab within 1 month prior to the randomization visit in either eye
* Study eye treatment with ITV anti-VEGF agents other than ranibizumab within 1 month prior to the randomization visit
* History of laser photocoagulation, Visudyne®, ITV corticosteroid injection, vitrectomy surgery, submacular surgery, device implantation, or other surgical intervention for AMD in the study eye
* Prior participation in a clinical trial involving anti-angiogenic drugs, other than ranibizumab, in either eye within 2 months of the randomization visit
* Subretinal hemorrhage in the study eye that involves the center of the fovea
* Subfoveal fibrosis, or atrophy in the study eye
* Choroidal neovascularization (CNV) in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Uncontrolled ocular hypertension or glaucoma in the study eye
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery in the study eye
* Uncontrolled blood pressure
* Uncontrolled atrial fibrillation within 3 months of informed consent
* History of myocardial infarction or stroke within the last 3 months prior to informed consent
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the Implant, that might affect interpretation of the results of the study or renders the participant at high risk of treatment complications
* Use of oral corticosteroids
* Current treatment for any active systemic infection
* Use of anticoagulants, anti-platelets (other than aspirin), or medications known to exert similar effects
* Active malignancy within 12 months of randomization
* History of allergy to fluorescein
* Previous participation in any non-ocular (systemic) disease studies of investigational drugs within 1 month preceding the informed consent (excluding vitamins and minerals)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- United States (50):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - The Retina Partners, Encino, California
  - Jacobs Retina center at the Shiley eye Institute UCSD, La Jolla, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - N CA Retina Vitreous Assoc, Mountain View, California
  - Retinal Consultants Med Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - UCSF; Ophthalmology, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Florida Eye Microsurgical Inst, Boynton Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Illinois Retina Associates, Joliet, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Johns Hopkins Med; Wilmer Eye Inst, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Vitreoretinal Surgery, Edina, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - University of New Mexico; School of Med, Albuquerque, New Mexico
  - Retina Assoc of Western NY, Rochester, New York
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Retina Northwest, Portland, Oregon
  - Oregon HSU; Casey Eye Institute, Portland, Oregon
  - Palmetto Retina Center, Florence, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Wagner Macula & Retina Center, Norfolk, Virginia

REFERENCES:
- [Derived] Campochiaro PA, Eichenbaum D, Chang MA, Clark WL, Graff JM, Le Pogam S, Cavichini Cordeiro M, Gune S, Rabena M, Singh N, Lin S, Callaway N. Interim Results of the Phase III Portal Extension Trial of the Port Delivery System with Ranibizumab in Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2025 Feb;9(2):144-155. doi: 10.1016/j.oret.2024.05.021. Epub 2024 Aug 30. PMID 39209113
- [Derived] Wykoff CC, Campochiaro PA, Pieramici DJ, Khanani AM, Gune S, Maia M, Kagedal M, Ding HT, Maass KF. Pharmacokinetics of the Port Delivery System with Ranibizumab in the Ladder Phase 2 Trial for Neovascular Age-Related Macular Degeneration. Ophthalmol Ther. 2022 Oct;11(5):1705-1717. doi: 10.1007/s40123-022-00532-9. Epub 2022 Jun 27. PMID 35759124
- [Derived] Awh CC, Barteselli G, Makadia S, Chang RT, Stewart JM, Wieland MR, Brassard R, Callaway NF, Gune S, Heatherton P, Malhotra V, Willis JR, Pieramici DJ. Management of Key Ocular Adverse Events in Patients Implanted with the Port Delivery System with Ranibizumab. Ophthalmol Retina. 2022 Nov;6(11):1028-1043. doi: 10.1016/j.oret.2022.05.011. Epub 2022 May 16. PMID 35589078
- [Derived] Yohe S, Maass KF, Horvath J, Rea J, Barteselli G, Ranade SV. In-vitro characterization of ranibizumab release from the Port Delivery System. J Control Release. 2022 May;345:101-107. doi: 10.1016/j.jconrel.2022.03.005. Epub 2022 Mar 4. PMID 35248647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with subfoveal neovascularization secondary to AMD diagnosed within 9 months and treated with ITV anti-VEGF agents were enrolled in the study. Written informed consent was obtained before initiation of any study-related procedures. A participant's screening occurred no sooner than 7 days following administration of the last ITV ranibizumab treatment to the study eye. The screening visit was followed by the randomization visit.
Period: Overall Study
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Started | 59 | 62 | 63 | 41
Completed | 51 | 56 | 56 | 36
Not Completed | 8 | 6 | 7 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 3 | 1 | 1 | 0
Not completed — Participant moved out of the area | 0 | 0 | 0 | 1
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg | Total
Number analyzed (Participants) | 59 | 62 | 63 | 41 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 9 | 7 | 31
  >=65 years | 51 | 55 | 54 | 34 | 194
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.6 (8.4) | 75.0 (8.5) | 73.8 (8.1) | 71.9 (8.8) | 74.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 42 | 28 | 146
  Male | 22 | 23 | 21 | 13 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 1 | 10
  Not Hispanic or Latino | 56 | 56 | 60 | 39 | 211
  Unknown or Not Reported | 0 | 3 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 58 | 61 | 60 | 41 | 220
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time Until a Participant First Requires the Implant Refill According to Protocol-Defined Refill Criteria
Description: Protocol-Defined Refill Criteria
  At 1 month after initial fill:
  * Decrease of ≥ 10 letters in BCVA at the current visit compared with the baseline BCVA, due to nAMD disease activity OR
  * Increase in CFT of ≥ 100 um at the current visit compared with the baseline CFT, due to nAMD disease activity OR
  * Presence of new macular hemorrhage, due to nAMD disease activity
  For subsequent assessments:
  * Increase in CFT of ≥ 75 μm on SD-OCT at the current visit compared with the average CFT over the last 2 available measurements, due to nAMD disease activity OR
  * Increase in CFT of ≥ 100 um from the lowest CFT measurement on study, due to nAMD disease activity OR
  * Decrease of ≥ 5 letters in BCVA at the current visit compared with the average BCVA over the last 2 available measurements, due to nAMD disease activity OR
  * Decrease of ≥ 10 letters from best recorded BCVA on study, due to nAMD disease activity OR
  * Presence of new macular hemorrhage, due to nAMD disease activity
Time Frame: Baseline up to approximately 38 months
Population: Efficacy Population defined as all participants who were randomly assigned to study treatment and received at least one study treatment, excluding 5 participants who were given surgery.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL
Number analyzed (Participants) | 58 | 62 | 59
Months | 8.7 [6.93 to 9.00] | 13.0 [11.76 to 24.61] | 15.8 [12.06 to 20.63]

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Averaged At Month 9 and 10
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. The minimum score possible is 0 and maximum possible is 100. A higher score represents better functioning.
Time Frame: Baseline, Months 9, 10
Population: Efficacy Population defined as all participants who were randomly assigned to study treatment and received at least one study treatment. Assessments are censored for PDS participants meeting the following situations:
  * At the time of an ITV anti-VEGF injection in study eye prior to Month 10.
  * Prohibited therapy other than oral corticosteroids more than 10 mg/day or any fellow eye treatment.
  * At the time of explant.
Measure: Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 58 | 62 | 59 | 41
Units on scale | -3.3 [-5.6 to -1.0] | -0.3 [-2.5 to 1.8] | 5.0 [2.8 to 7.2] | 3.2 [0.6 to 5.8]

3. Secondary Outcome: Change From Baseline in BCVA Over Time
Description: as for outcome 2
Time Frame: Baseline up to Month 10
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 58 | 62 | 59 | 41
Units on scale
  Month 1: number analyzed (Participants) | 58 | 62 | 58 | 41
  Month 1 | -6.6 [-11.0 to -2.3] | -4.7 [-8.8 to -0.6] | -4.9 [-9.1 to -0.6] | 2.4 [-2.6 to 7.5]
  Month 2: number analyzed (Participants) | 58 | 60 | 58 | 41
  Month 2 | -2.4 [-4.3 to -0.6] | -1.4 [-3.2 to 0.4] | 1.6 [-0.2 to 3.5] | 2.0 [-0.2 to 4.2]
  Month 3: number analyzed (Participants) | 57 | 60 | 58 | 40
  Month 3 | -0.7 [-2.4 to 1.0] | -0.6 [-2.2 to 1.0] | 2.4 [0.8 to 4.1] | 2.7 [0.7 to 4.7]
  Month 4: number analyzed (Participants) | 58 | 60 | 59 | 41
  Month 4 | -1.4 [-3.4 to 0.7] | -1.1 [-3.0 to 0.8] | 3.1 [1.1 to 5.1] | 1.9 [-0.4 to 4.3]
  Month 5: number analyzed (Participants) | 58 | 61 | 58 | 41
  Month 5 | -1.3 [-3.4 to 0.8] | -0.6 [-2.5 to 1.4] | 3.8 [1.8 to 5.8] | 3.0 [0.6 to 5.3]
  Month 6: number analyzed (Participants) | 58 | 61 | 58 | 41
  Month 6 | -0.4 [-3.0 to 2.3] | -1.7 [-4.3 to 0.8] | 3.8 [1.2 to 6.4] | 2.7 [-0.4 to 5.7]
  Month 7: number analyzed (Participants) | 58 | 61 | 58 | 40
  Month 7 | -0.9 [-3.2 to 1.4] | -1.8 [-4.0 to 0.3] | 3.9 [1.7 to 6.1] | 3.5 [0.9 to 6.1]
  Month 8: number analyzed (Participants) | 57 | 60 | 57 | 40
  Month 8 | -2.4 [-4.7 to -0.1] | -1.2 [-3.3 to 1.0] | 4.0 [1.8 to 6.2] | 3.3 [0.7 to 5.9]
  Month 9: number analyzed (Participants) | 57 | 59 | 56 | 37
  Month 9 | -3.3 [-5.7 to -0.9] | -0.5 [-2.7 to 1.7] | 5.0 [2.7 to 7.3] | 3.9 [1.1 to 6.6]
  Month 10: number analyzed (Participants) | 58 | 62 | 58 | 37
  Month 10 | -3.3 [-5.7 to -1.0] | -0.2 [-2.4 to 2.0] | 5.1 [2.8 to 7.3] | 2.5 [-0.2 to 5.2]

4. Secondary Outcome: Adjusted Average Change From Baseline in BCVA Over Time (MMRM Analysis)
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. The minimum score possible is 0 and maximum possible is 100. A higher score represents better functioning. Here, the adjusted mean from MMRM analysis is presented).
Time Frame: Baseline up to Month 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 45 | 60 | 55 | 37
Units on scale | -7.5 (74.0) | -8.5 (59.1) | 29.7 (54.7) | 21.3 (65.1)

5. Secondary Outcome: Change From Baseline in Central Foveal Thickness (CFT) Over Time as Assessed on Spectral Domain-Optical Coherence Tomography (SD-OCT)
Description: Central foveal thickness (CFT) is defined as the retinal thickness in the center of the fovea
Time Frame: Baseline up to Month 9
Population: Efficacy Population defined as all participants who received at least one study treatment. Here, "Number of Participants analyzed" indicates Number of Participants Included in MMRM Analysis. Assessments are censored for PDS participants meeting the following situations:
  * At the time of an ITV anti-VEGF injection in study eye prior to Month 10.
  * Prohibited therapy other than oral corticosteroids more than 10 mg/day or any fellow eye treatment.
  * At the time of explant.
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 58 | 62 | 59 | 41
microns
  Month 1: number analyzed (Participants) | 52 | 59 | 55 | 41
  Month 1 | 16.5 [4.1 to 29.0] | 7.2 [-4.5 to 18.9] | -2.9 [-15.1 to 9.2] | 2.5 [-11.7 to 16.7]
  Month 2: number analyzed (Participants) | 56 | 59 | 55 | 41
  Month 2 | 19.8 [6.9 to 32.7] | 11.9 [-0.3 to 24.1] | -1.8 [-14.5 to 10.9] | 1.5 [-13.3 to 16.4]
  Month 3: number analyzed (Participants) | 56 | 57 | 57 | 39
  Month 3 | 24.9 [11.5 to 38.3] | 7.3 [-5.5 to 20.0] | 6.4 [-6.8 to 19.6] | -7.3 [-22.9 to 8.3]
  Month 4: number analyzed (Participants) | 54 | 60 | 57 | 41
  Month 4 | 31.0 [15.8 to 46.1] | 4.1 [-10.3 to 18.5] | 1.9 [-13.2 to 16.9] | -1.7 [-19.2 to 15.9]
  Month 5: number analyzed (Participants) | 58 | 60 | 57 | 41
  Month 5 | 30.9 [16.1 to 45.7] | 0.4 [-13.6 to 14.5] | 8.0 [-6.7 to 22.9] | 4.0 [-13.0 to 21.1]
  Month 6: number analyzed (Participants) | 58 | 59 | 58 | 41
  Month 6 | 31.9 [15.6 to 48.1] | 2.1 [-13.1 to 17.3] | 5.9 [-10.0 to 21.7] | -2.0 [-20.4 to 16.4]
  Month 7: number analyzed (Participants) | 57 | 59 | 53 | 40
  Month 7 | 39.9 [25.6 to 54.3] | 0.7 [-12.5 to 14.0] | -4.3 [-18.3 to 9.6] | -9.8 [-25.9 to 6.3]
  Month 8: number analyzed (Participants) | 56 | 56 | 56 | 38
  Month 8 | 42.8 [26.4 to 59.1] | 3.1 [-12.1 to 18.3] | 5.1 [-10.6 to 20.8] | -2.4 [-20.8 to 16.1]
  Month 9 | 54.8 [37.1 to 72.4] | -0.7 [-16.9 to 15.5] | -1.7 [-18.5 to 15.1] | -6.3 [-26.1 to 13.4]

6. Secondary Outcome: Number of Implant Clogging at Month 9
Description: Removed implants identified as meeting serum PK criteria for possible clogging were assessed via lab-based investigation (in vitro drug release testing) to determine whether there was any implant clogging.
Time Frame: Month 9
Population: Efficacy Population defined as all participants who were randomly assigned to study treatment and received at least one study treatment.
Measure: Number; unit: Participants
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL
Number analyzed (Participants) | 58 | 62 | 59
Participants | 0 | 0 | 0

7. Secondary Outcome: Observed Maximum Serum Concentration (Cmax) of Ranibizumab
Description: The serum pharmacokinetics of ranibizumab were characterized by estimating Cmax between dose intervals. Estimates for these parameters were tabulated and summarized by descriptive statistics.
Time Frame: Predose (0 hour) on Day 1 up to 38 months
Population: PK Population with exclusion (randomized participants who had received at least one study drug administration and provided at least one serum and/or aqueous PK sample for determination of ranibizumab concentration excluding participants who had prior intravitreal bevacizumab, received fellow eye ranibizumab treatment, and/or received supplemental intravitreal ranibizumab)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 16 | 25 | 27 | 0
pg/mL
  Interval following implant insertion before first refill | 105.52 (258.0) | 220.87 (46.4) | 1080.69 (272.5) |
  All Dose Intervals | 91.47 (187.2) | 297.61 (115.2) | 1131.01 (256.6) |

8. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing to Last Observation (AUClast) of Ranibizumab
Description: AUCLast is defined as area under the concentration-time curve from dosing (implant or refill) to last observation before next refill or exiting the study. The serum pharmacokinetics of ranibizumab were characterized by estimating AUC between dose intervals. Estimates for these parameters were tabulated and summarized by descriptive statistics.
Time Frame: Predose (0 hour) on Day 1 up to approximately 38 months (detailed timeframe is provided in description field)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙day/mL
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 16 | 25 | 27 | 0
ng∙day/mL
  Interval following implant insertion before first refill | 5.89 (225.1) | 28.39 (107.6) | 90.83 (64.7) |
  All Dose Intervals | 3.43 (176.8) | 22.93 (96.9) | 66.12 (71.4) |

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of Ranibizumab
Description: The serum pharmacokinetics of ranibizumab were characterized by estimating Tmax between dose intervals. Estimates for these parameters were tabulated and summarized by descriptive statistics.
Time Frame: Predose (0 hour) on Day 1 up to 38 months
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 16 | 25 | 27 | 0
days
  Interval following implant insertion before first refill | 11.45 [0 to 688.1] | 12.87 [0 to 86.0] | 29.01 [0.8 to 180.3] |
  All Dose Intervals | 4.87 [0 to 688.1] | 6.71 [0 to 91.1] | 6.97 [0.8 to 180.3] |

10. Secondary Outcome: Terminal Half-Life (t1/2) of Ranibizumab
Description: The serum pharmacokinetics of ranibizumab were characterized by estimating t1/2 between dose intervals. Estimates for these parameters were tabulated and summarized by descriptive statistics.
Time Frame: Predose (0 hour) on Day 1 up to 38 months
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 16 | 25 | 27 | 0
days
  Interval following implant insertion before first refill: number analyzed (Participants) | 11 | 23 | 24 | 0
  Interval following implant insertion before first refill | 168.20 (163.3) | 88.30 (46.7) | 119.07 (128.4) |
  All Dose Intervals | 162.36 (129.3) | 118.87 (76.2) | 143.87 (171.4) |

11. Secondary Outcome: Observed Steady-State Serum Concentration at the End of a Dosing Interval (Ctrough) of Ranibizumab
Time Frame: Predose (0 hour) on Day 1 up to 38 months
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 16 | 25 | 27 | 0
pg/mL
  Interval following implant insertion before first refill: number analyzed (Participants) | 7 | 9 | 12 | 0
  Interval following implant insertion before first refill | 14.96 (76.4) | 61.64 (95.8) | 129.63 (149.2) |
  All Dose Intervals | 11.58 (65.7) | 105.07 (77.4) | 62.19 (345.2) |

12. Secondary Outcome: Number of Participants With Ocular and Non-Ocular Adverse Events (AEs) and Serious AEs (SAEs)
Time Frame: Baseline up to approximately Month 38
Population: Safety analyses were based on the Safety Population which was composed of participants receiving at least one study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Ranibizumab PD All Participants: Participants had the Implant (prefilled with approximately 20 μL either the 10 mg/mL [approximately 0.2 mg dose], 40 mg/mL [approximately 0.8 mg dose], or 100 mg/mL formulation [approximately 2-mg dose] of ranibizumab) surgically inserted in the study eye at the Day 1 visit following their randomization visit. Starting at the Month 1 visit, participants were evaluated monthly for the need for Implant refill with the 10 mg/mL, 40 mg/mL, or 100 mg/mL formulations of ranibizumab according to their randomization as per protocol-specified refill criteria.
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Ranibizumab PD All Participants | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 58 | 62 | 59 | 179 | 41
Participants
  Participants with ocular SAEs in study eye | 7 | 6 | 4 | 17 | 0
  Participants with ocular AEs in study eye | 56 | 58 | 52 | 166 | 26
  Participants with non-ocular SAEs | 8 | 16 | 13 | 37 | 4
  Participants with non-ocular AEs | 46 | 52 | 52 | 150 | 36

13. Secondary Outcome: Percentage of Participants With Positive Serum Antibodies to Ranibizumab
Time Frame: Baseline up to 38 months
Population: Safety analyses were based on the Safety Population which was composed of participants receiving at least one study treatment. Here, number of analyzed participants represents number of participants from whom samples were collected and analyzed. Baseline evaluable participant is a participant with an ADA assay result from a baseline sample(s). Post-baseline evaluable participant is a participant with an ADA assay result from at least one post-baseline sample.
Measure: Number; unit: Percentage of Participants
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Ranibizumab PD All Participants | Intravitreal Injection With Ranibizumab 0.5mg
Number analyzed (Participants) | 58 | 62 | 59 | 179 | 41
Percentage of Participants
  Participants with a positive sample at time of entry into the study (Baseline): number analyzed (Participants) | 58 | 60 | 59 | 177 | 39
  Participants with a positive sample at time of entry into the study (Baseline) | 10.3 | 5.0 | 5.1 | 6.8 | 0
  Participants positive for Treatment Emergent ADA (Post-baseline) | 6.9 | 14.5 | 15.3 | 12.3 | 14.6

ADVERSE EVENTS:
Time Frame: Baseline up to approximately Month 38
Description: Number of events includes all occurrences. Table summary includes adverse events that started or worsened (for existing condition) on or after the date of first study treatment during the study.
Arm/Group | Port Delivery System With Ranibizumab 10mg/mL | Port Delivery System With Ranibizumab 40mg/mL | Port Delivery System With Ranibizumab 100mg/mL | Intravitreal Injection With Ranibizumab 0.5mg
All-Cause Mortality (participants affected / at risk) | 1/58 | 2/62 | 1/59 | 1/41
Serious Adverse Events (participants affected / at risk) | 14/58 | 19/62 | 17/59 | 4/41
Other Adverse Events (participants affected / at risk) | 57/58 | 59/62 | 58/59 | 35/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Port Delivery System With Ranibizumab 10mg/mL (N=58) | Port Delivery System With Ranibizumab 40mg/mL (N=62) | Port Delivery System With Ranibizumab 100mg/mL (N=59) | Intravitreal Injection With Ranibizumab 0.5mg (N=41)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL EROSION (Eye disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
HYPOTONY OF EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL TEAR (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
RETINOPATHY PROLIFERATIVE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHEGMATOGENOUS RETINAL DETACHMENT (Eye disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
TRACTIONAL RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
VITREOUS HAEMORRHAGE (Eye disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOPHTHALMITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 4 (6) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL FILTERING BLEB LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVAL RETRACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPHAEMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ILIOTIBIAL BAND SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OCULAR PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND SECRETION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Port Delivery System With Ranibizumab 10mg/mL (N=58) | Port Delivery System With Ranibizumab 40mg/mL (N=62) | Port Delivery System With Ranibizumab 100mg/mL (N=59) | Intravitreal Injection With Ranibizumab 0.5mg (N=41)
ANTERIOR CHAMBER CELL (Eye disorders) | 1 (1) | 2 (2) | 6 (6) | 0 (0)
ANTERIOR CHAMBER FLARE (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
BLEPHARITIS (Eye disorders) | 1 (1) | 1 (1) | 3 (8) | 1 (1)
CATARACT (Eye disorders) | 3 (4) | 5 (8) | 12 (16) | 5 (7)
CATARACT CORTICAL (Eye disorders) | 3 (3) | 2 (3) | 0 (0) | 3 (5)
CATARACT NUCLEAR (Eye disorders) | 3 (3) | 3 (3) | 2 (3) | 1 (2)
CHOROIDAL DETACHMENT (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
CONJUNCTIVAL BLEB (Eye disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 41 (53) | 44 (54) | 37 (38) | 8 (11)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 18 (20) | 13 (14) | 14 (16) | 0 (0)
CONJUNCTIVAL OEDEMA (Eye disorders) | 6 (7) | 6 (6) | 1 (1) | 0 (0)
CORNEAL OEDEMA (Eye disorders) | 6 (6) | 3 (3) | 4 (4) | 0 (0)
DERMATOCHALASIS (Eye disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
DIPLOPIA (Eye disorders) | 3 (4) | 3 (4) | 1 (2) | 1 (2)
DRY EYE (Eye disorders) | 7 (10) | 2 (3) | 5 (7) | 1 (2)
EYE DISCHARGE (Eye disorders) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
EYE IRRITATION (Eye disorders) | 9 (9) | 7 (9) | 7 (7) | 2 (3)
EYE PAIN (Eye disorders) | 12 (16) | 12 (15) | 15 (18) | 5 (7)
EYELID OEDEMA (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
EYELID PTOSIS (Eye disorders) | 3 (3) | 2 (2) | 4 (4) | 1 (1)
EYELIDS PRURITUS (Eye disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 4 (6) | 7 (7) | 7 (8) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
IRITIS (Eye disorders) | 8 (9) | 13 (14) | 7 (7) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 3 (4) | 2 (3) | 0 (0) | 0 (0)
MACULAR DEGENERATION (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
NEOVASCULAR AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 8 (8) | 10 (10) | 10 (12) | 3 (3)
OCULAR HYPERAEMIA (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 4 (6) | 5 (7) | 5 (7) | 5 (6)
PUNCTATE KERATITIS (Eye disorders) | 5 (7) | 3 (4) | 2 (3) | 1 (1)
RETINAL HAEMORRHAGE (Eye disorders) | 6 (7) | 6 (11) | 5 (5) | 1 (1)
VISION BLURRED (Eye disorders) | 8 (11) | 3 (8) | 5 (6) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (3) | 3 (3) | 3 (5) | 0 (0)
VITREOUS DETACHMENT (Eye disorders) | 7 (7) | 6 (8) | 4 (6) | 7 (9)
VITREOUS DISORDER (Eye disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
VITREOUS FLOATERS (Eye disorders) | 13 (13) | 9 (13) | 12 (15) | 4 (5)
VITREOUS HAEMORRHAGE (Eye disorders) | 4 (4) | 5 (6) | 4 (6) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 5 (6) | 4 (5) | 4 (4) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
BRONCHITIS (Infections and infestations) | 3 (3) | 9 (9) | 4 (4) | 5 (6)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
EAR INFECTION (Infections and infestations) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
HORDEOLUM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
INFLUENZA (Infections and infestations) | 5 (5) | 1 (1) | 4 (4) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 12 (17) | 8 (15) | 9 (11) | 6 (9)
SINUSITIS (Infections and infestations) | 2 (2) | 5 (7) | 9 (11) | 7 (9)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 6 (6) | 3 (3) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 5 (6) | 10 (17) | 6 (9) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 5 (6) | 1 (1)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 4 (6) | 0 (0)
HYPHAEMA (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 5 (5) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 4 (5) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
INTRAOCULAR PRESSURE DECREASED (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 8 (14) | 3 (3) | 6 (8) | 3 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (7) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 6 (6) | 4 (4)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 4 (6) | 3 (4) | 2 (2)
HEADACHE (Nervous system disorders) | 9 (10) | 8 (9) | 11 (11) | 1 (1)
HYPERTONIC BLADDER (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 2 (2) | 2 (2)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
HYPERTENSION (Vascular disorders) | 5 (5) | 2 (2) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT02510794/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT02510794/SAP_001.pdf